CLINICAL TRIAL: NCT02706197
Title: A Single-Institutional, Phase 1 Trial of Repeated Oxygen Measurements in Subcutaneous Tumors by Electron Paramagnetic Resonance (EPR) Oximetry Using an Implantable Oxygen Sensor (OxyChip)
Brief Title: Oxygen Measurements in Subcutaneous Tumors by EPR Oximetry Using OxyChip
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study halted prematurely but potentially will resume
Sponsor: Periannan Kuppusamy (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Periannan Kuppusamy, Scientific Director, Dartmouth-Hitchcock Medical Center
Organization: Dartmouth-Hitchcock Medical Center (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 28499 D14007; P01CA190193 (NIH)
Record Dates: First submitted 2016-02-26; First posted 2016-03-11 (Estimated); Results first posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Neoplasms, Benign; Neoplasms, Malignant
Keywords: Electron Paramagnetic Resonance; Hypoxia; OxyChip
MeSH Terms: conditions — Neoplasms; Hypoxia

STUDY DESIGN:
Intervention Model Description: There are two parallel arms of the study; however, the first 6 patients must be in the arm whose tumor will receive no therapy prior to surgical resection. If there are no safety issues, then both arms are open.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- IA No treatment except standard-of-care (SOC) surgery (Experimental): Placement of OxyChip will be through a minimally invasive procedure (needle injection) and removal will be at the time of surgical resection. In Phase IA, patients will not have any cancer therapy prior to removal of the OxyChip and duration of implantation is typically less than 4 weeks but may be up to 52 weeks.
  Interventions: Device: OxyChip
- IB SOC adjuvant therapy and SOC surgery (Experimental): Placement of OxyChip will be through a minimally invasive procedure (needle injection) and removal will be at the time of surgical resection. In Phase IB, patients will have standard of care neoadjuvant chemotherapy or pre-operative radiation therapy during the time that the OxyChip is within the tumor, which is typically 6 weeks but may be up to 52 weeks.
  Interventions: Device: OxyChip

INTERVENTIONS:
Device: OxyChip — The OxyChip is an investigational device to assess oxygen level in tissues, when measured with Electron Paramagnetic Resonance (EPR).
  Other Names: implantable oxygen sensor

SUMMARY:
Tumors with low oxygen levels are associated with poor prognosis and resistance to standard radiotherapy or systemic therapies. The ability to make repeated oxygen measurements in tumors could be used to help select the most effective treatment or the best timing to start therapies. The purpose of this study is to ascertain the safety and feasibility of using an implantable oxygen sensor, known as the OxyChip, to make oxygen measurements in tumors using EPR oximetry, a technique related to magnetic resonance imaging (MRI).

DETAILED DESCRIPTION:
This is an early feasibility Phase I clinical trial for safety. The total enrollment for this study is 60 patients (30 per phase). The study is split in a phase IA (short duration of implantation with no other cancer therapy planned prior to excision) and a phase IB (duration of implantation for up to 52 weeks while receiving neoadjuvant radiation therapy or systemic therapy prior to surgical excision), as described below.

The initial 6 patients will have the OxyChip placed for a short duration (up to 4 weeks) after which the OxyChip will be removed when the tumor mass is resected, prior to delivery of any further therapies. After the successful implantation, removal, and evaluation of the OxyChip in the first 6 Phase IA patients, enrollment will be opened to an additional 24 Phase IA patients and to 6 Phase IB patients who will either receive neoadjuvant radiotherapy or systemic therapy (chemotherapy, biologic therapy, or endocrine therapy) while the OxyChip is in place. After the successful implantation, removal, and evaluation of the OxyChip in the first 3 Phase IB patients receiving radiation therapy or systemic therapy, enrollment will be opened to an additional 24 Phase IB patients. Up to five oxygen measurements per week will be made during the course of radiation or systemic therapy. The OxyChips will be removed at surgery. Patients receiving radiation or systemic therapy will be evaluated at least weekly for assessment with respect to any adverse events for the primary objective and oximetry measurements will be taken periodically at least one day after implantation and up to its removal at the planned tumor excision to assess the secondary objective. Following resection, the tissue surrounding the OxyChip will be examined for any adverse events for the primary objective. For the exploratory objectives, the tissue will also be examined for biomarkers associated with hypoxia or growth.

ELIGIBILITY:
Inclusion Criteria:

1. Phase IA: Any tumor identified by imaging or physical exam to be accessable to OxyChip implantation and measurements and that is going to receive surgical resection with intent to remove the entire tumor. The tumor must be sufficiently large to accommodate the OxyChip.
2. Phase IB: Any biopsy-proven malignancy expected to undergo neoadjuvant chemotherapy or radiotherapy prior to resection. The tumor must be sufficiently large to accommodate the OxyChip.
3. The tumor must be within 3 cm of the surface of the skin or mucosa.
4. Age ≥18 years old.
5. Subject must be capable of giving informed consent.
6. Anticipated time between implantation and planned surgical excision of at least three days.
7. Tumors must be > 2.5 cm in minimum diameter to be eligible.

Exclusion Criteria:

1. Pregnant women or women of childbearing potential without adequate contraception. Contraception, which can include abstinence, is required from the first day of the last menstrual period until the removal of the OxyChip.
2. Receipt of concurrent chemotherapy and radiotherapy, or planned sequential chemotherapy and radiotherapy, prior to resection (Phase IB),
3. Receipt of Avastin, or other angiogenesis inhibitors, during the study.
4. Prior radiotherapy to the site of implantation.
5. Having other implanted (not removable) devices that generate electrical artifacts or that could be altered by the EPR magnetic field, such as cardiac pacemakers or defibrillators.
6. Concurrent enrollment in any clinical research study, in the absence of cancer recurrence, in which the other study can reasonably be anticipated to have the potential for causing adverse events that would affect our primary endpoint of assessing the safety of the OxyChip device. If a study is not felt to impact the evaluation of adverse events in this trial then the patient will be eligible for concurrent enrollment. In the presence of confirmed clinical recurrence after initial cancer therapy (and after removal of OxyChip) during the year-long follow up stipulated in the protocol, patients will be eligible for all clinical trials as deemed appropriate by the treating oncologist.
7. Patient platelet blood count < 50,000/l of blood, and absolute neutrophil count < 1,000/l of blood. Laboratory values must be obtained at least 3 months prior to implantation of the OxyChip.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-12-31 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip E Schaner, M.D., Ph.D., Principal Investigator — Dartmouth-Hitchcock Medical Center; Periannan Kuppusamy, Ph.D., Principal Investigator — Dartmouth College
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brizel DM, Dodge RK, Clough RW, Dewhirst MW. Oxygenation of head and neck cancer: changes during radiotherapy and impact on treatment outcome. Radiother Oncol. 1999 Nov;53(2):113-7. doi: 10.1016/s0167-8140(99)00102-4. PMID 10665787
- [Background] Vaupel P, Thews O, Hoeckel M. Treatment resistance of solid tumors: role of hypoxia and anemia. Med Oncol. 2001;18(4):243-59. doi: 10.1385/MO:18:4:243. PMID 11918451
- [Background] Swartz HM, Walczak T. Developing in vivo EPR oximetry for clinical use. Adv Exp Med Biol. 1998;454:243-52. doi: 10.1007/978-1-4615-4863-8_29. PMID 9889898
- [Background] Doll CM, Milosevic M, Pintilie M, Hill RP, Fyles AW. Estimating hypoxic status in human tumors: a simulation using Eppendorf oxygen probe data in cervical cancer patients. Int J Radiat Oncol Biol Phys. 2003 Apr 1;55(5):1239-46. doi: 10.1016/s0360-3016(02)04474-7. PMID 12654433
- [Background] Gagel B, Piroth M, Pinkawa M, Reinartz P, Zimny M, Kaiser HJ, Stanzel S, Asadpour B, Demirel C, Hamacher K, Coenen HH, Scholbach T, Maneschi P, DiMartino E, Eble MJ. pO polarography, contrast enhanced color duplex sonography (CDS), [18F] fluoromisonidazole and [18F] fluorodeoxyglucose positron emission tomography: validated methods for the evaluation of therapy-relevant tumor oxygenation or only bricks in the puzzle of tumor hypoxia? BMC Cancer. 2007 Jun 28;7:113. doi: 10.1186/1471-2407-7-113. PMID 17598907
- [Background] Vaupel P, Mayer A. Hypoxia in cancer: significance and impact on clinical outcome. Cancer Metastasis Rev. 2007 Jun;26(2):225-39. doi: 10.1007/s10555-007-9055-1. PMID 17440684
- [Background] Cosse JP, Michiels C. Tumour hypoxia affects the responsiveness of cancer cells to chemotherapy and promotes cancer progression. Anticancer Agents Med Chem. 2008 Oct;8(7):790-7. doi: 10.2174/187152008785914798. PMID 18855580
- [Background] Shannon AM, Bouchier-Hayes DJ, Condron CM, Toomey D. Tumour hypoxia, chemotherapeutic resistance and hypoxia-related therapies. Cancer Treat Rev. 2003 Aug;29(4):297-307. doi: 10.1016/s0305-7372(03)00003-3. PMID 12927570
- [Background] Tatum JL, Kelloff GJ, Gillies RJ, Arbeit JM, Brown JM, Chao KS, Chapman JD, Eckelman WC, Fyles AW, Giaccia AJ, Hill RP, Koch CJ, Krishna MC, Krohn KA, Lewis JS, Mason RP, Melillo G, Padhani AR, Powis G, Rajendran JG, Reba R, Robinson SP, Semenza GL, Swartz HM, Vaupel P, Yang D, Croft B, Hoffman J, Liu G, Stone H, Sullivan D. Hypoxia: importance in tumor biology, noninvasive measurement by imaging, and value of its measurement in the management of cancer therapy. Int J Radiat Biol. 2006 Oct;82(10):699-757. doi: 10.1080/09553000601002324. PMID 17118889
- [Background] Vaupel P. Hypoxia and aggressive tumor phenotype: implications for therapy and prognosis. Oncologist. 2008;13 Suppl 3:21-6. doi: 10.1634/theoncologist.13-S3-21. PMID 18458121
- [Background] Cardenas-Navia LI, Yu D, Braun RD, Brizel DM, Secomb TW, Dewhirst MW. Tumor-dependent kinetics of partial pressure of oxygen fluctuations during air and oxygen breathing. Cancer Res. 2004 Sep 1;64(17):6010-7. doi: 10.1158/0008-5472.CAN-03-0947. PMID 15342381
- [Background] Cardenas-Navia LI, Mace D, Richardson RA, Wilson DF, Shan S, Dewhirst MW. The pervasive presence of fluctuating oxygenation in tumors. Cancer Res. 2008 Jul 15;68(14):5812-9. doi: 10.1158/0008-5472.CAN-07-6387. PMID 18632635
- [Background] O'Hara JA, Blumenthal RD, Grinberg OY, Demidenko E, Grinberg S, Wilmot CM, Taylor AM, Goldenberg DM, Swartz HM. Response to radioimmunotherapy correlates with tumor pO2 measured by EPR oximetry in human tumor xenografts. Radiat Res. 2001 Mar;155(3):466-73. doi: 10.1667/0033-7587(2001)155[0466:rtrcwt]2.0.co;2. PMID 11182798
- [Background] O'Hara JA, Goda F, Dunn JF, Swartz HM. Potential for EPR oximetry to guide treatment planning for tumors. Adv Exp Med Biol. 1997;411:233-42. doi: 10.1007/978-1-4615-5865-1_28. No abstract available. PMID 9269432
- [Background] Pandian RP, Dolgos M, Marginean C, Woodward PM, Hammel PC, Manoharan PT, Kuppusamy P. Molecular packing and magnetic properties of lithium naphthalocyanine crystals: hollow channels enabling permeability and paramagnetic sensitivity to molecular oxygen. J Mater Chem. 2009;19(24):4138-4147. doi: 10.1039/b901886g. PMID 19809598
- [Background] Pandian RP, Parinandi NL, Ilangovan G, Zweier JL, Kuppusamy P. Novel particulate spin probe for targeted determination of oxygen in cells and tissues. Free Radic Biol Med. 2003 Nov 1;35(9):1138-48. doi: 10.1016/s0891-5849(03)00496-9. PMID 14572616
- [Background] Meenakshisundaram G, Eteshola E, Pandian RP, Bratasz A, Selvendiran K, Lee SC, Krishna MC, Swartz HM, Kuppusamy P. Oxygen sensitivity and biocompatibility of an implantable paramagnetic probe for repeated measurements of tissue oxygenation. Biomed Microdevices. 2009 Aug;11(4):817-26. doi: 10.1007/s10544-009-9298-4. PMID 19319683
- [Background] Meenakshisundaram G, Pandian RP, Eteshola E, Lee SC, Kuppusamy P. A paramagnetic implant containing lithium naphthalocyanine microcrystals for high-resolution biological oximetry. J Magn Reson. 2010 Mar;203(1):185-9. doi: 10.1016/j.jmr.2009.11.016. Epub 2009 Nov 26. PMID 20006529
- [Derived] Schaner PE, Pettus JR, Flood AB, Williams BB, Jarvis LA, Chen EY, Pastel DA, Zuurbier RA, diFlorio-Alexander RM, Swartz HM, Kuppusamy P. OxyChip Implantation and Subsequent Electron Paramagnetic Resonance Oximetry in Human Tumors Is Safe and Feasible: First Experience in 24 Patients. Front Oncol. 2020 Oct 27;10:572060. doi: 10.3389/fonc.2020.572060. eCollection 2020. PMID 33194670

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 25 patients were recruited starting from 12/31/2015 to 9/26/2018 in the radiation Oncology Clinic of Dartmouth Hospital.
Pre-assignment Details: Out of the 25 enrolled, one participant had signed consent, but withdrew consent prior to any measurement activities.
Period: Overall Study
Arm/Group | IA No Treatment Except Standard-of-care (SOC) Surgery | IB SOC Adjuvant Therapy and SOC Surgery
Started | 18 | 6
Completed | 18 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IA No Treatment Except Standard-of-care (SOC) Surgery | IB SOC Adjuvant Therapy and SOC Surgery | Total
Number analyzed (Participants) | 18 | 6 | 24
Age, Continuous [Mean (Full Range); unit: Years] | 64.1 [42 to 83] | 53.5 [23 to 70] | 61.4 [23 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 12 | 1 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 17 | 6 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 18 | 6 | 24

OUTCOME MEASURES:

1. Primary Outcome: Safety of OxyChip by Recording of Adverse Events as Measured by Histological Signs of Tissue Reaction and Inflammation
Description: This is a safety study to demonstrate that the OxyChip will be well-tolerated with minimal risk for complications. All tumors will be excised with the OxyChip in place, and histology will be analyzed for signs of tissue reaction and inflammation adjacent to the OxyChip. pathologic findings associated with the OxyChip are reported.
Time Frame: From time of implantation procedure to 2 weeks after removal of OxyChip, up to 18 weeks
Population: The OxyChip could not be found for two participants. The chip was presumed to be lost at the time of surgery for one participant and presumed lost prior to surgery due to rapidly progressive tumor necrosis.
Measure: Count of Participants; unit: Participants
Arm/Group | IA No Treatment Except Standard-of-care (SOC) Surgery | IB SOC Adjuvant Therapy and SOC Surgery
Number analyzed (Participants) | 16 | 6
Participants
  Focal disrupted tissue at edge of tumor with mild nonspecific chronic inflammation | 1 | 0
  Focal fibrosis, macrophages, and apparent tumor cavitation | 1 | 0
  Focal organizing fat necrosis | 1 | 0
  Mild macrophage and foreign body type giant cell reaction at OxyChip site | 1 | 0
  Mild macrophage predominant chronic inflammatory reaction at needle site | 1 | 0
  Minimal fat necrosis, macrophage infiltrate immediately surrounding the OxyChip | 1 | 0
  Minor focal hemorrhage seen adjacent to the deep margin. Very focal collection of macrophages. | 1 | 0
  Minor hemorrhage at site of injection | 1 | 0
  Tumor necrosis and mild hemorrhage immediately adjacent to injection site | 1 | 0
  Tumor necrosis near chip site. | 1 | 0
  No histologic response seen | 6 | 5
  Focal fibrosis, a few macrophages adjacent | 0 | 1

2. Primary Outcome: Safety of OxyChip by Recording of Adverse Events (Allergic Reaction, Infection, Hemorrhage, Skin Erosion Over the Device, Device Breakage or Malfunction)
Description: This is a safety study to demonstrate that the implantation procedure, the OxyChip and any subsequent oxygen measurements will be well-tolerated with minimal risk for complications.
Time Frame: From time of implantation procedure to 2 weeks after removal of OxyChip
Measure: Count of Participants; unit: Participants
Arm/Group | IA No Treatment Except Standard-of-care (SOC) Surgery | IB SOC Adjuvant Therapy and SOC Surgery
Number analyzed (Participants) | 18 | 6
Participants
  Discomfort at surgical site | 1 | 0
  Mild discomfort and bleeding from implantation procedure. Bruising from implantation needle | 0 | 1
  Mild discomfort from implantation | 0 | 1
  Minimal bleeding associated with implantation. Mild bruising at needle insertion site | 1 | 0
  Minor bleeding asociated w implantation. Minor bruising needle ins site. Mild discomfort of L breast | 0 | 1
  Minor bleeding from implantation needle | 5 | 2
  Minor bleeding from implantation needle. Mild bruising. | 2 | 0
  Minor bruising associated with implantation site | 1 | 0
  No Adverse Events Recorded | 5 | 1
  Pain and minor bleeding from implantation needle | 1 | 0
  Pruritis | 1 | 0
  Pruritis, scalp | 1 | 0

3. Secondary Outcome: Measurement of Tumor Partial Pressure of Oxygen (pO2) Levels Using the OxyChip Sensor and EPR Oximetry
Description: This study will also determine the feasibility of repeated measurements of pO2 in tumors using the OxyChip and EPR oximetry. Tumor pO2 values will be reported in millimeters of mercury (mmHg).
  Two types of measurements (Data) were made: (i) Baseline tumor pO2 values in patients breathing room air during the first up to 10 min period; and (ii) Hyperoxygenation pO2 values at the end of patients breathing 100% oxygen gas for up to 10 min. The hyperoxygenation was administered immediately following the baseline (room-air breathing) measurements.
Time Frame: From time of implantation procedure to time of OxyChip removal; an average of 2 weeks for Phase IA and up to 4 months for Phase IB
Population: For Arm 1A, 4 subjects were not measured. For Arm 1B, 4 subjects were not measured.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | IA No Treatment Except Standard-of-care (SOC) Surgery | IB SOC Adjuvant Therapy and SOC Surgery
Number analyzed (Participants) | 14 | 2
mmHg
  Baseline pO2 data | 17.1 (17.4) | 18.8 (8.8)
  Hyperoxygen pO2 data measured immediately following baseline pO2 data | 41.7 (35.7) | 42.7 (38.6)

4. Secondary Outcome: The Time Required to Complete EPR Oximetry Measurements
Description: This study will also determine the feasibility of repeated measurements of oxygen in tumors using the OxyChip and EPR oximetry. We will determine the workflow and time required for each daily oxygen measurement. The measurement time, averaged over multiple measurements on each patient, will be reported as less than or greater than one hour.
Time Frame: From time of preparing the patient for EPR measurement, for example placement of the patient on the bed, attaching the resonator, to completion of the EPR measurements, for example, detaching the resonator and removing the patient off the bed.
Population: One subject from IA had Oxychip presumed lost at time of surgery. 4 subjects from each group were not able to be measured.
Measure: Count of Participants; unit: Participants
Arm/Group | IA No Treatment Except Standard-of-care (SOC) Surgery | IB SOC Adjuvant Therapy and SOC Surgery
Number analyzed (Participants) | 14 | 2
Participants
  Less than 1 Hour | 14 | 2
  Greater than 1 Hour | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events will be evaluated at each study visit, from baseline through 12 months following implantation.
Description: Events were evaluated for associated toxicity using the Common Terminology Criteria for Adverse Events (CTCAE);
Arm/Group | IA No Treatment Except Standard-of-care (SOC) Surgery | IB SOC Adjuvant Therapy and SOC Surgery
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/6
Other Adverse Events (participants affected / at risk) | 13/18 | 5/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IA No Treatment Except Standard-of-care (SOC) Surgery (N=18) | IB SOC Adjuvant Therapy and SOC Surgery (N=6)
Minor Bleeding (Surgical and medical procedures) | 10 (10) | 4 (4)
Pain/Discomfort (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Bruising (Injury, poisoning and procedural complications) | 4 (4) | 2 (2)
Pruritis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan: Study Protocol and Statistical Analysis Plan (2018-07-10): https://cdn.clinicaltrials.gov/large-docs/97/NCT02706197/Prot_SAP_000.pdf